CLINICAL TRIAL: NCT00033215
Title: A Phase 1 Study of S-3304 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0110P1416
Record Dates: First submitted 2002-04-09; First posted 2002-04-10 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Solid Tumors
Keywords: neovascularization; matrix metalloproteinases; antiangiogenesis; type IV collagenases
MeSH Terms: conditions — Neovascularization, Pathologic | interventions — S 3304

STUDY DESIGN:
Intervention Model Description: Four dose levels were evaluated sequentially in separate groups of 6 to 8 patients: 1,600 mg/d (800 mg BID, Dose Level1 (DL1)), 3,200 mg/d (1,600 mg BID, DL2), 4,800 mg/d (2,400 mg BID, DL3), and 6,400 mg/d (3,200 mg BID, DL4). There was no intrapatient dose escalation.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: S-3304

SUMMARY:
To determine the maximum tolerated dose and safety profile of S-3304 in patients with biopsy accessible cancer who have failed previous therapy or to whom no standard therapies are available. To determine the pharmacokinetic profile of S-3304 in this patient population

ELIGIBILITY:
Inclusion criteria:

* Biopsy proven diagnosis of solid tumor(s) with biopsy accessible lesion(s)
* Must be able to tolerate oral medication Exclusion criteria
* Patients with other serious illnesses
* Patients who are receiving treatments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2001-11 (Actual); Primary Completion 2003-02-13 (Actual); Study Completion 2003-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado Hospital, Denver, Colorado
  - H. Lee Moffitt Concer Center and Research Institute, Tampa, Florida
  - Roswell Park Cancer Center, Buffalo, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Result] Chiappori AA, Eckhardt SG, Bukowski R, Sullivan DM, Ikeda M, Yano Y, Yamada-Sawada T, Kambayashi Y, Tanaka K, Javle MM, Mekhail T, O'bryant CL, Creaven PJ. A phase I pharmacokinetic and pharmacodynamic study of s-3304, a novel matrix metalloproteinase inhibitor, in patients with advanced and refractory solid tumors. Clin Cancer Res. 2007 Apr 1;13(7):2091-9. doi: 10.1158/1078-0432.CCR-06-1586. PMID 17404091